CLINICAL TRIAL: NCT04422431
Title: A Phase 2, Single-arm Pathologist-blinded 48-week Study Using Liver Biopsy Specimens to Assess Copper Concentration and Histopathologic Changes in ALXN1840-treated Patients With Wilson Disease Followed by an up to 48-weeks Extension Period
Brief Title: Copper Concentration & Histopathologic Changes in Liver Biopsy in Participants With Wilson Disease Treated With ALXN1840
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALXN1840-WD-205; 2019-003711-60 (EudraCT Number)
Record Dates: First submitted 2020-05-22; First posted 2020-06-09 (Actual); Results first posted 2023-07-03 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Wilson Disease
Keywords: Copper; ALXN1840; Histology; Liver Biopsy
MeSH Terms: conditions — Hepatolenticular Degeneration | interventions — tetrathiomolybdate

STUDY DESIGN:
Masking Description: This study is only pathologist-blinded for the assessments of liver histology samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ALXN1840 (Experimental): Participants will receive ALXN1840.
  Interventions: Drug: Bis-Choline Tetrathiomolybdate

INTERVENTIONS:
Drug: Bis-Choline Tetrathiomolybdate — Participants will be initiated at 15 milligrams once daily, then the dose will be increased to 30 milligrams once daily at Week 6.
  Other Names: ALXN1840

SUMMARY:
The main objective of the study is to evaluate the change in liver copper (Cu) concentration following 48 weeks of treatment with ALXN1840 in adult participants with Wilson Disease (WD) who have been previously treated for at least 1 year with standard of care (that is, trientine, penicillamine, or zinc). In the Treatment Period, efficacy and safety of ALXN1840 will be assessed at Week 48.

DETAILED DESCRIPTION:
Participants who complete the 48-week Treatment Period will be offered the opportunity to continue their treatment in a 48-week Extension Period that will offer additional time for evaluation of long-term efficacy and safety of ALXN1840. There will be no liver biopsies during the Extension Period.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of WD by Leipzig Criteria ≥ 4 or by historical test results.
2. Continuous treatment for WD with penicillamine, trientine or zinc for at least 1 year prior to screening.
3. Body mass index < 30 kilograms/meter squared.
4. Able to cooperate with a percutaneous liver biopsy.
5. Willing and able to follow protocol-specified contraception requirements.
6. Capable of giving signed informed consent.

Exclusion Criteria:

1. Decompensated cirrhosis or Model for End Stage Liver Disease score > 13.
2. Modified Nazer score > 7.
3. Clinically significant gastrointestinal bleed within past 3 months.
4. Alanine aminotransferase > 2 × upper limit of normal.
5. History of bleeding abnormality or known coagulopathy, including platelet count < 100,000, and international normalized ratio for prothrombin time ≥ 1.5.
6. Participant unwilling to accept blood products, if required.
7. Marked neurological disease requiring either nasogastric feeding tube or intensive inpatient medical care.
8. Hemoglobin less than lower limit of the reference range for age and sex.
9. Participants in renal failure, defined as in end-stage renal disease on dialysis (chronic kidney disease 5) or creatinine clearance < 30 milliliters/minute.
10. Lymphoma, leukemia, or any malignancy within the past 5 years.
11. Current or chronic history of liver disease not associated with WD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2022-05-21 (Actual); Study Completion 2023-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene S. Swenson, MD, PhD, Study Director — Alexion Pharmaceuticals, Inc.
Locations (12):
- United States (3):
  - Research Site, Sacramento, California
  - Research Site, Ann Arbor, Michigan
  - Research Site, Dallas, Texas
- Research Site, Toronto, Ontario, Canada
- Research Site, Århus N, Denmark
- Research Site, Grafton, New Zealand
- Russia (2):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- Research Site, Singapore, Singapore
- Spain (2):
  - Research Site, Barcelona
  - Research Site, Valencia
- Research Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ALXN1840-WD-205&attachmentIdentifier=165b7460-1a66-4ad7-9b5f-7bb17c7d363e&fileName=ALXN1840-WD-205_CSR_Synopsis_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- ALXN1840: Participants received ALXN1840 orally in the 48-week Treatment Period. Participants who completed the 48-week Treatment Period and agreed to enter a 48-week Extension Period, continued to receive ALXN1840. Participants who did not enter the Extension Period discontinued dosing at Week 48, and had a final study visit for safety follow-up at Week 52.
Period: Treatment Period (48 Weeks)
Arm/Group | ALXN1840
Started | 31
Received at Least 1 Dose of Study Drug | 31
Completed | 26
Not Completed | 5
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 1
Not completed — Other than specified | 1
Period: Extension Period (48 Weeks)
Arm/Group | ALXN1840
Started | 25 (1 participant completed Treatment Period but did not enter the Extension Period.)
Received at Least 1 Dose of Study Drug | 25
Completed | 21
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1
Not completed — Other than specified | 2

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set in the Treatment Period included all participants who received at least 1 dose of study drug in the Treatment Period and had at least a Baseline liver copper (Cu) value evaluable.
Arm/Group | ALXN1840
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.9 (13.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 19
  Race: Asian | 6
  Race: Other | 3
  Race: Unknown | 1
Liver Cu Concentration [Mean (Standard Deviation); unit: micrograms (μg)/gram (g)] | 511.2 (361.85)
Hepatic Collagen Content [Mean (Standard Deviation); unit: percentage of collagen] | 10.2993 (6.81501)
Alpha-Smooth Muscle Actin (a-SMA) Content [Mean (Standard Deviation); unit: percentage of a-SMA] | 5.3134 (3.25982)
Hepatic Fat Content [Mean (Standard Deviation); unit: percentage of fat] | 1.5815 (2.60491)
Non-alcoholic Fatty Liver Disease (NAFLD) Activity Score (NAS) Total Score [Mean (Standard Deviation); unit: units on a scale] — Inflammation was quantified by the NAS total score. The score is defined as the unweighted sum of the scores for steatosis (0 [minimal] to 3 [severe]), lobular inflammation (0 [none] to 3 [>4 foci / 200x field]), and hepatocellular ballooning (0 [none] to 2 [many]), thus ranging from 0 (no inflammation) to 8 (severe inflammation), with higher scores indicating more severe disease.
  units on a scale | 1.2 (1.45)
Molybdenum (Mo) in Liver Biopsy Specimen [Mean (Standard Deviation); unit: μg/g] | 4.1591 (4.43552)
Clinical Global Impression-Severity (CGI-S) Scale Score [Mean (Standard Deviation); unit: units on a scale] — The CGI-S is a 7-point scale clinician assessment. Participants were assessed on severity of illness at the time of rating/assessment as follows: 1 = normal, not at all ill; 2 = borderline ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; or 7 = extremely ill. Higher scores indicated worsening of disease.
  units on a scale | 2.3 (1.26)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Liver Cu Concentration at Week 48 (Treatment Period)
Description: Liver biopsy samples were taken for the assessment of liver Cu concentration. Multiple imputation was used to impute missing data at Week 48 due to any reason based on Baseline values.
Time Frame: Baseline, Week 48 (Treatment Period)
Population: The Full Analysis Set in the Treatment Period included all participants who received at least 1 dose of study drug in the Treatment Period and had at least a Baseline liver Cu value evaluable.
Measure: Mean (Standard Error); unit: μg/g
Arm/Group | ALXN1840
Number analyzed (Participants) | 29
μg/g | 92.8 (56.34)
Statistical Analysis 1: Comparison: ALXN1840; Test type: Other; p = 0.1002, t-test, 2 sided

2. Secondary Outcome: Number of Participants With Change From Baseline in Nonalcoholic Steatohepatitis Clinical Research Network (NASH CRN) Fibrosis Stage at Week 48 (Treatment Period)
Description: Fibrosis from histology was evaluated by NASH CRN Fibrosis Stage, which was scaled from 0 to 4 stages where Score 0: None; Score 1: Perisinusoidal or periportal - 1a - mild, zone 3, perisinusoidal; Score 1: Perisinusoidal or periportal - 1b - moderate, zone 3, perisinusoidal; Score 1: Perisinusoidal or periportal - 1c - portal/periportal; Score 2: Both perisinusoidal and portal/periportal; Score 3: Bridging fibrosis; and Score 4: Cirrhosis. Higher scores indicated greater fibrosis.
Time Frame: Baseline, Week 48 (Treatment Period)
Population: The Full Analysis Set in the Treatment Period included all participants who received at least 1 dose of study drug in the Treatment Period and had at least a Baseline liver Cu value evaluable. 'Number analyzed' signifies participants evaluable at specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | ALXN1840
Number analyzed (Participants) | 29
Participants
  Baseline: Score 0 | 7
  Baseline: Score 1a | 1
  Baseline: Score 1b | 0
  Baseline: Score 1c | 7
  Baseline: Score 2 | 3
  Baseline: Score 3 | 8
  Baseline: Score 4 | 2
  Baseline: Not evaluable | 1
  Week 48: number analyzed (Participants) | 24
  Week 48: Score 0 | 5
  Week 48: Score 1a | 0
  Week 48: Score 1b | 0
  Week 48: Score 1c | 6
  Week 48: Score 2 | 6
  Week 48: Score 3 | 7
  Week 48: Score 4 | 0
  Week 48: Not evaluable | 0

3. Secondary Outcome: Number of Participants With Change From Baseline in Metavir Fibrosis Score at Week 48 (Treatment Period)
Description: Fibrosis from histology was evaluated by Metavir Fibrosis Score, which was ranged from 0 to 4 where Score 0: No fibrosis; Score 1: Stellate enlargement of portal tract but without septa formation; Score 2: Enlargement of portal tract with rare septa formation; Score 3: Numerous septa without cirrhosis; and Score 4: Cirrhosis. Higher scores indicated greater fibrosis.
Time Frame: Baseline, Week 48 (Treatment Period)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | ALXN1840
Number analyzed (Participants) | 29
Participants
  Baseline: Score 0 | 8
  Baseline: Score 1 | 7
  Baseline: Score 2 | 4
  Baseline: Score 3 | 7
  Baseline: Score 4 | 2
  Baseline: Not evaluable | 1
  Week 48: number analyzed (Participants) | 24
  Week 48: Score 0 | 5
  Week 48: Score 1 | 4
  Week 48: Score 2 | 8
  Week 48: Score 3 | 7
  Week 48: Score 4 | 0
  Week 48: Not evaluable | 0

4. Secondary Outcome: Number of Participants With Change From Baseline in Ishak Fibrosis Score at Week 48 (Treatment Period)
Description: Fibrosis from histology was evaluated by Ishak Fibrosis Score, which was ranged from 0 to 6 where Score 0: No fibrosis; Score 1: Fibrous expansion of some portal areas, with or without short fibrous septa; Score 2: Fibrous expansion of most portal areas, with or without short fibrous septa; Score 3: Fibrous expansion of most portal areas with occasional portal to portal (P-P) bridging; and Score 4: Fibrous expansion of portal areas with marked bridging (P-P) as well as portal central (P-C); Score 5: Marked bridging (P-P and/or P-C) with occasional nodules (incomplete cirrhosis); and Score 6: Cirrhosis, probable or definite. Higher scores indicated greater fibrosis.
Time Frame: Baseline, Week 48 (Treatment Period)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | ALXN1840
Number analyzed (Participants) | 29
Participants
  Baseline: Score 0 | 8
  Baseline: Score 1 | 6
  Baseline: Score 2 | 2
  Baseline: Score 3 | 9
  Baseline: Score 4 | 1
  Baseline: Score 5 | 1
  Baseline: Score 6 | 1
  Baseline: Not evaluable | 1
  Week 48: number analyzed (Participants) | 24
  Week 48: Score 0 | 5
  Week 48: Score 1 | 4
  Week 48: Score 2 | 4
  Week 48: Score 3 | 8
  Week 48: Score 4 | 3
  Week 48: Score 5 | 0
  Week 48: Score 6 | 0
  Week 48: Not evaluable | 0

5. Secondary Outcome: Change From Baseline in Hepatic Collagen Content at Week 48 (Treatment Period)
Description: Fibrosis from histology was evaluated by morphometric quantification of hepatic collagen content.
Time Frame: Baseline, Week 48 (Treatment Period)
Population: The Full Analysis Set in the Treatment Period included all participants who received at least 1 dose of study drug in the Treatment Period and had at least a Baseline liver Cu value evaluable. 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percentage of collagen
Arm/Group | ALXN1840
Number analyzed (Participants) | 24
percentage of collagen | 8.5445 (15.54224)

6. Secondary Outcome: Change From Baseline in a-SMA Content at Week 48 (Treatment Period)
Description: Fibrosis from histology was evaluated by morphometric quantification of hepatic a-SMA content.
Time Frame: Baseline, Week 48 (Treatment Period)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentage of a-SMA
Arm/Group | ALXN1840
Number analyzed (Participants) | 24
percentage of a-SMA | 1.6002 (5.47274)

7. Secondary Outcome: Number of Participants With Change From Baseline in NAS Steatosis Grading Score at Week 48 (Treatment Period)
Description: Steatosis from histology was evaluated by the steatosis component of the NAS, which was ranged from 0 to 3 where Score 0: < 5% (minimal); Score 1: 5 - 33% (mild); Score 2: 34 - 66% (moderate); and Score 3: > 66% (severe). Higher scores indicated greater steatosis.
Time Frame: Baseline, Week 48 (Treatment Period)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | ALXN1840
Number analyzed (Participants) | 29
Participants
  Baseline: Score 0 | 19
  Baseline: Score 1 | 6
  Baseline: Score 2 | 3
  Baseline: Score 3 | 1
  Week 48: number analyzed (Participants) | 24
  Week 48: Score 0 | 15
  Week 48: Score 1 | 6
  Week 48: Score 2 | 2
  Week 48: Score 3 | 1

8. Secondary Outcome: Change From Baseline in Hepatic Fat Content at Week 48 (Treatment Period)
Description: Steatosis from histology was evaluated by morphometric quantification of hepatic fat content.
Time Frame: Baseline, Week 48 (Treatment Period)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentage of fat
Arm/Group | ALXN1840
Number analyzed (Participants) | 24
percentage of fat | -0.2504 (2.19263)

9. Secondary Outcome: Change From Baseline in NAS Total Score at Week 48 (Treatment Period)
Description: Inflammation was quantified by the NAS total score. The score is defined as the unweighted sum of the scores for steatosis (0 [minimal] to 3 [severe]), lobular inflammation (0 [none] to 3 [>4 foci / 200x field]), and hepatocellular ballooning (0 [none] to 2 [many]), thus ranging from 0 (no inflammation) to 8 (severe inflammation), with higher scores indicating more severe disease.
Time Frame: Baseline, Week 48 (Treatment Period)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ALXN1840
Number analyzed (Participants) | 24
units on a scale | 0.1 (1.69)

10. Secondary Outcome: Treatment Period: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An SAE was an AE that met at least 1 of the following criteria: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization for the AE, persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, congenital anomaly/birth defect (in the child of a participant who was exposed to the study drug), important medical event or reaction. The TEAEs were AEs with onset on or after the first study drug dose. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Day 1 (Treatment Period) up to Week 48 (Treatment Period)
Population: Safety Analysis Set in the Treatment Period included all participants who received at least 1 dose of treatment in the Treatment Period.
Measure: Count of Participants; unit: Participants
Arm/Group | ALXN1840
Number analyzed (Participants) | 31
Participants | 30

11. Secondary Outcome: Extension Period: Number of Participants With TEAEs
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An SAE was an AE that met at least 1 of the following criteria: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization for the AE, persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, congenital anomaly/birth defect (in the child of a participant who was exposed to the study drug), important medical event or reaction. The TEAEs were AEs with onset on or after the first study drug dose. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Day 1 (Extension Period) up Week 52 (Extension Period)
Population: Safety Analysis Set in the Extension Period included all participants who received at least 1 dose of ALXN1840 in the Extension Period.
Measure: Count of Participants; unit: Participants
Arm/Group | ALXN1840
Number analyzed (Participants) | 25
Participants | 24

12. Secondary Outcome: Treatment Period: Predose Trough Plasma Total Mo Concentration
Time Frame: Predose up to 4 hours postdose at Week 6 (Day 43) and Week 36 (Day 253)
Population: Pharmacokinetic (PK) Analysis Set in the Treatment Period included all participants who received at least 1 dose of treatment in the Treatment Period and had evaluable PK data for total Mo and/or plasma ultrafiltrate (PUF) Mo (as surrogate measure for ALXN1840 PK) in plasma in the Treatment Period. 'Overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: nanograms (ng)/milliliter (mL)
Arm/Group | ALXN1840
Number analyzed (Participants) | 29
nanograms (ng)/milliliter (mL)
  Week 6 | 174.39 (113.824)
  Week 36: number analyzed (Participants) | 28
  Week 36 | 131.19 (103.359)

13. Secondary Outcome: Treatment Period: Predose Trough Plasma Total PUF Mo Concentration
Time Frame: Predose up to 4 hours postdose at Week 6 (Day 43) and Week 36 (Day 253)
Population: PK Analysis Set in the Treatment Period included all participants who received at least 1 dose of treatment in the Treatment Period and had evaluable PK data for total Mo and/or PUF Mo (as surrogate measure for ALXN1840 PK) in plasma in the Treatment Period. 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ALXN1840
Number analyzed (Participants) | 28
ng/mL
  Week 6 | 5.888 (2.0176)
  Week 36 | 7.843 (6.0564)

14. Secondary Outcome: Change From Baseline in Mo in Liver Biopsy Specimen at Week 48 (Treatment Period)
Time Frame: Baseline, Week 48 (Treatment Period)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: μg/g
Arm/Group | ALXN1840
Number analyzed (Participants) | 24
μg/g | 69.6976 (43.02655)

15. Secondary Outcome: Clinical Global Impression-Improvement (CGI-I) Scale Score at Week 48 (Treatment Period)
Description: The CGI-I is a 7-point scale clinician assessment where 1= very much improved; 2 = much improved; 3 = minimally improved; 4 = no change; 5 = minimally worse; 6 = much worse; or 7 = very much worse. Higher scores indicated worsening of disease.
Time Frame: Week 48 (Treatment Period)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ALXN1840
Number analyzed (Participants) | 25
units on a scale | 3.1 (1.26)

16. Secondary Outcome: Change From Baseline in CGI-S Scale Score at Week 48 (Treatment Period)
Description: The CGI-S is a 7-point scale clinician assessment. Participants were assessed on severity of illness at the time of rating/assessment as follows: 1 = normal, not at all ill; 2 = borderline ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; or 7 = extremely ill. Higher scores indicated worsening of disease.
Time Frame: Baseline, Week 48 (Treatment Period)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ALXN1840
Number analyzed (Participants) | 25
units on a scale | -0.4 (1.50)

ADVERSE EVENTS:
Time Frame: Day 1 (Treatment Period) up to Week 52 (Extension Period) (up to a total of approximately 100 weeks)
Description: All-cause mortality is reported for all enrolled participants in both periods. Serious and other adverse events are reported in the Safety Analysis Set in the Treatment Period, which included all participants who received at least 1 dose of treatment in the Treatment Period, and for the Safety Analysis Set in the Extension Period, which included all participants who received at least 1 dose of ALXN1840 in the Extension Period.
Groups:
- Treatment Period: ALXN1840: Participants received ALXN1840 orally in the 48-week Treatment Period.
- Extension Period: ALXN1840: Participants who completed the 48-week Treatment Period and agreed to enter a 48-week Extension Period, continued to receive ALXN1840.
Arm/Group | Treatment Period: ALXN1840 | Extension Period: ALXN1840
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/25
Serious Adverse Events (participants affected / at risk) | 3/31 | 2/25
Other Adverse Events (participants affected / at risk) | 30/31 | 24/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Period: ALXN1840 (N=31) | Extension Period: ALXN1840 (N=25)
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Bence Jones proteinuria (Renal and urinary disorders) | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Treatment Period: ALXN1840 (N=31) | Extension Period: ALXN1840 (N=25)
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 2 | 2
Chalazion (Eye disorders) | 1 | 1
Vision blurred (Eye disorders) | 1 | 0
Vitreous detachment (Eye disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 6 | 6
Abdominal discomfort (Gastrointestinal disorders) | 2 | 3
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Oral pain (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 2
Faeces discoloured (Gastrointestinal disorders) | 1 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 2
Haemorrhoids thrombosed (Gastrointestinal disorders) | 1 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 1
Toothache (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 5 | 3
Fatigue (General disorders) | 4 | 2
Asthenia (General disorders) | 2 | 2
Chills (General disorders) | 2 | 0
Feeling abnormal (General disorders) | 2 | 2
Generalised oedema (General disorders) | 1 | 1
Pain (General disorders) | 1 | 0
Temperature intolerance (General disorders) | 1 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 2 | 2
Seasonal allergy (Immune system disorders) | 2 | 2
Immunisation reaction (Immune system disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 5 | 8
COVID-19 (Infections and infestations) | 4 | 10
Kidney infection (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 4
Urinary tract infection (Infections and infestations) | 2 | 1
Bacterial vaginosis (Infections and infestations) | 1 | 0
Conjunctivitis (Infections and infestations) | 1 | 1
Dermatophytosis (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 1 | 0
Furuncle (Infections and infestations) | 1 | 0
Gingivitis (Infections and infestations) | 1 | 1
Helicobacter infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1
Paronychia (Infections and infestations) | 1 | 1
Post procedural sepsis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Incision site pain (Injury, poisoning and procedural complications) | 1 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 1
Post procedural fever (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 | 0
Post procedural hypotension (Injury, poisoning and procedural complications) | 1 | 0
Post procedural swelling (Injury, poisoning and procedural complications) | 1 | 0
Post vaccination syndrome (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 1
Alanine aminotransferase increased (Investigations) | 8 | 8
Gamma-glutamyltransferase increased (Investigations) | 8 | 7
Blood alkaline phosphatase increased (Investigations) | 4 | 4
Hepatic enzyme increased (Investigations) | 4 | 2
Aspartate aminotransferase increased (Investigations) | 3 | 2
Blood creatine phosphokinase increased (Investigations) | 3 | 4
Transaminases increased (Investigations) | 3 | 2
Blood bilirubin increased (Investigations) | 2 | 1
Liver function test increased (Investigations) | 2 | 2
Alanine aminotransferase abnormal (Investigations) | 1 | 1
Blood albumin decreased (Investigations) | 1 | 0
Blood folate decreased (Investigations) | 1 | 1
Creatinine renal clearance decreased (Investigations) | 1 | 0
Creatinine renal clearance increased (Investigations) | 1 | 1
Protein urine present (Investigations) | 1 | 0
Prothrombin time prolonged (Investigations) | 1 | 0
Urobilinogen urine increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 1
Weight increased (Investigations) | 1 | 1
White blood cell count decreased (Investigations) | 1 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 | 3
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Greater trochanteric pain syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Headache (Nervous system disorders) | 7 | 6
Lethargy (Nervous system disorders) | 3 | 2
Dizziness (Nervous system disorders) | 2 | 2
Presyncope (Nervous system disorders) | 2 | 2
Tremor (Nervous system disorders) | 2 | 1
Balance disorder (Nervous system disorders) | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 2
Anxiety disorder (Psychiatric disorders) | 1 | 1
Depressed mood (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 2
Personality disorder (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Glycosuria (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 1
Breast mass (Reproductive system and breast disorders) | 1 | 1
Breast tenderness (Reproductive system and breast disorders) | 1 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1/11 | 1/9 — The N at risk for this adverse event has been adjusted to the number of females in the respective study periods as it is a sex-specific event.
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1/11 | 0/9 — The N at risk for this adverse event has been adjusted to the number of females in the respective study periods as it is a sex-specific event.
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1/11 | 2/9 — The N at risk for this adverse event has been adjusted to the number of females in the respective study periods as it is a sex-specific event.
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 2
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0
Idiopathic guttate hypomelanosis (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 2
Myopia (Eye disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1
Neck injury (Injury, poisoning and procedural complications) | 0 | 1
Procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 2
Viral upper respiratory tract infection (Infections and infestations) | 0 | 2
Bacteriuria (Infections and infestations) | 0 | 1
Urine analysis abnormal (Investigations) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Serotonin syndrome (Nervous system disorders) | 0 | 1
Influenza like illness (General disorders) | 0 | 1
Swelling (General disorders) | 0 | 1
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 | 1
Back disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Mixed anxiety and depressive disorder (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Ingrown hair (Skin and subcutaneous tissue disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-05-27): https://cdn.clinicaltrials.gov/large-docs/31/NCT04422431/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-22): https://cdn.clinicaltrials.gov/large-docs/31/NCT04422431/SAP_001.pdf